CLINICAL TRIAL: NCT00713063
Title: Behavioral Exercise Intervention for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0603-01; 5K23DA019950 (NIH)
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Nicotine Dependence
Keywords: smoking cessation; exercise; physical activity; health education
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Motor Activity; Health Education | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 12-week moderate intensity behavioral exercise intervention (MIBE) AND a 12-week standard smoking cessation program (including transdermal nicotine patch)
  Interventions: Behavioral: aerobic exercise
- 2 (Active Comparator): 12-week health education control (HEC) AND a 12-week standard smoking cessation program (including transdermal nicotine patch).
  Interventions: Behavioral: Health Education Control

INTERVENTIONS:
Behavioral: aerobic exercise — 12-week moderate intensity behavioral exercise intervention (MIBE) AND a 12-week standard smoking cessation program (including transdermal nicotine patch)
  Arms: 1
Behavioral: Health Education Control — 12-week health education control (HEC) AND a 12-week standard smoking cessation program (including transdermal nicotine patch).
  Arms: 2

SUMMARY:
The purpose of this study is to test the effect of a moderate-intensity aerobic exercise intervention for smokers interested in quitting smoking. We expect that this project will contribute much needed knowledge about the role of aerobic exercise in smoking cessation. If the efficacy of moderate-intensity, aerobic exercise for smoking can be established, smokers may have a valuable adjunct to more traditional smoking cessation approaches.

ELIGIBILITY:
Inclusion Criteria:

1. are between 18 and 65 years of age
2. are current smokers (i.e., smoking at least 10 cigarettes per day)
3. are sedentary, i.e., have not participated regularly in aerobic physical exercise (for at least 20 minutes per day, 3 days per week) for the past six months.

Exclusion Criteria:

1. current DSM-IV Axis I psychiatric disorder as assessed by SCID-NP
2. Substance abuse or dependence (excluding nicotine dependence) within the past 6 months
3. lifetime DSM-IV diagnosis of a bipolar disorder as assessed by the SCID-NP
4. lifetime history of a psychotic disorder or current psychotic symptoms as assessed by the SCID-NP
5. current suicidality or homicidality
6. marked organic impairment
7. physical disabilities or medical problems (such as a history of diabetes, hypertension, seizure disorder, coronary heart disease, valvular heart disease, and pulmonary disease) or use of medications (such as beta blockers) that would prevent or hinder participation in a program of moderate intensity exercise
8. current pregnancy of intent to become pregnant during the next 12 weeks, and i) current use of any pharmacotherapy, including transdermal nicotine replacement, for smoking cessation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Self-reported smoking abstinence via Timeline Followback (TLFB) | 12-months
Biochemically verified smoking abstinence via carbon monoxide and saliva cotinine | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ana Abrantes, PhD, Principal Investigator — Butler Hospital